CLINICAL TRIAL: NCT02904070
Title: Interest of Placental Alpha-microglobulin-1 Detection Test to Assess Risk of Premature Delivery in Reunion Island
Acronym: PARTOSURE-OI
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 2013/CHU/07
Record Dates: First submitted 2016-09-08; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Premature Delivery
Keywords: Threat of
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Threat of premature delivery (Experimental): * Perform detection test of Placental Alpha-Microglobulin-1, fetal Fibronectin and phosphorylated Insulin-like Growth Factor Binding Protein-1ph by vaginal swabbing;
  * Collection of clinical data, laboratory data and treatment of obstetric care in the delivery room during childbirth for all included subjects
  Interventions: Device: Vaginal swabbing

INTERVENTIONS:
Device: Vaginal swabbing

SUMMARY:
Prematurity is the leading cause of mortality and perinatal morbidity. Despite the many preventive measures and use of tocolytic therapy, the incidence of premature births has not decreased in recent decades. In 2010 the preterm birth rate (single child, born alive) was still 5.5% in France and 11% in the population of Reunion. In 50% of cases, premature birth is related to spontaneous premature labor layout without rupture of amniotic membranes, called threat of premature birth.The threat of premature birth, defined by the combination of cervical modifications and regular and painful uterine contractions from 22 weeks of amenorrhea and 36 weeks of amenorrhea + 6days, is the major cause of hospitalization in pathological pregnancies services. But all threat of premature delivery situations do not cause premature delivery. In our service, only 30% of patients hospitalized for threat of premature delivery give birth prematurely in accordance with published international data. The diagnosis of threat of premature delivery is difficult and it is still not possible to differentiate a "false labour" of a "real labour".

Currently the diagnosis of threat of premature delivery in routine is based on the combination of vaginal examination, the ultrasound, cervical length, but this strategy lacks specificity.

In absence of prognostic tool for predicting more reliably the risk of premature delivery in situation of threat of premature delivery, the medical cares are maximalist.: hospitalization, conducting paraclinical investigations, prescription of tocolytics treatments and conducting antenatal corticotherapy. it seems particularly necessary to identify more efficient prognostic criteria that the clinic and ultrasound for judging the severity of threat of premature delivery in other words to predict the risk of premature delivery to adapt and adjust the care of patients after diagnosis of threat of premature delivery.

ELIGIBILITY:
Inclusion Criteria:

* All patients received in programmed or emergency consultation;
* Pregnant, between 24 weeks of amenorrhea and 33 weeks of amenorrhea + 6 days;
* With painful regular uterine contractions confirmed by monitoring;
* Patient affiliated to a social security scheme;
* Informed consent signed by patient if adult or by legal representant for minor subjects

Exclusion Criteria:

* cervical cerclage placement;
* proved vaginal infection and/or vaginal ongoing treatment;

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Efficient predictivity for premature delivery assessed by Placental Alpha-microglobulin-1 detection test compared with the cervical length | Childbirth
  Occurrence of premature delivery within 7 days of diagnosis depending on the positive / negative status for the Placental Alpha-microglobulin-1 detection test versus cervical length

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa BENASSI, MD, Principal Investigator — CHU de La Réunion
Locations (1):
- CHU de La Réunion - site Nord, Saint-Denis, Reunion Island, France

IPD SHARING:
Plan to Share IPD: No